CLINICAL TRIAL: NCT06408493
Title: Peer-led Digital Health Lifestyle Intervention for a Low Income Community at Risk for Cardiovascular Diseases (MYCardio-PEER)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University Malaysia (Other)
Collaborators: Ministry of Higher Education, Malaysia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36440
Record Dates: First submitted 2024-03-18; First posted 2024-05-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Primary Prevention of Cardiovascular Diseases
Keywords: Peer-led; Primary prevention; Cardiovascular diseases; Digital health; Lifestyle intervention; Peer support; Community
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will attend the 8-weeks MYCardio-PEER program with their peer leaders, supplemented with face-to-face components.
  Interventions: Behavioral: MYCardio-PEER
- Control (No Intervention): Participants will receive printed documents with standard tips on dietary and lifestyle management for CVD.

INTERVENTIONS:
Behavioral: MYCardio-PEER — MYCardio-PEER participants will attend an 8-weeks intervention program delivered over the social networking application. Bite-sized videos and infographic posters on healthy diet and lifestyle for primary prevention of CVD will be delivered weekly, supplemented by interactive peer-group activities to encourage behavior change.
  Arms: Intervention

SUMMARY:
The goal of this interventional study is to develop and assess the effectiveness of a peer-led digital health program (MYCardio-PEER) for primary prevention of cardiovascular disease (CVD) in a low-income community at-risk of CVD.

The main questions it aims to answer are:

* Is MYCardio-PEER effective in improving knowledge, lifestyle behaviors and CVD biomarkers of a low-income community at-risk for CVD?
* Is there an association between MYCardio-PEER participants' adherence and satisfaction, with effectiveness and sustainability of the program?

Participants will attend the 8-weeks MYCardio-PEER program with their peer leaders, supplemented with face-to-face components. Participants will then be followed up for another 12 weeks, during which peer leaders and researchers will have minimal contact with the participants. Participants who have been allocated into the control group will receive printed documents with standard tips on dietary and lifestyle management for CVD, where they will be encouraged to maintain regular calorie intake and expenditure and perform regular exercise.

ELIGIBILITY:
Inclusion Criteria:

* Mentally sound man/woman of at least 30 years old
* Monthly household income of less than RM3,710 or receiving government aid for low-income community
* Literate with a fair command of the Malay language
* Have mobile device connected to the Internet
* Willing to attend 8 weeks of intervention and be followed up for another 12 weeks during the maintenance phase.
* Have been confirmed to have a moderate or high risk for CVD based on the Framingham General CVD Risk Score

Exclusion Criteria:

* Pregnant, lactating or intend to become pregnant during the study period.
* Any other pre-existing conditions or severe complications that could compromise the ability to adhere to the study program.
* Enrolled in other studies.

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Framingham Risk Score for Cardiovascular Disease Risk | 20 weeks
  The score is based on a person's age, sex, blood pressure, cholesterol levels, smoking status, and diabetes status. The calculated score will be converted into 10-year risk percentage whereby the higher the percentage means higher cardiovascular disease risk.

SECONDARY OUTCOMES:
Blood pressure | 20 weeks
  The blood pressure will be measured in mmHg. Blood pressure more than 140/90 mmHg is considered high blood pressure.
Total cholesterol level | 20 weeks
  Total cholesterol will be measured in mmol/L. Total cholesterol more than 5.2 mmol/L is considered high.
High-density lipoprotein cholesterol (HDL-C) level | 20 weeks
  High-density lipoprotein cholesterol (HDL-C) will be measured in mmol/L. The healthy cut-off points of HDL-C in male is more than 1.0 mmol/L and in female more than 1.3 mmol/L.
Low-density lipoprotein cholesterol (LDL-C) level | 20 weeks
  Low-density lipoprotein cholesterol (LDL-C) will be measured in mmol/L. The healthy cut-off point of LDL-C is less than 2.6 mmol/L.
Triglycerides level | 20 weeks
  Triglycerides level will be measured in mmol/L. The healthy cut-off point of triglycerides level is less than 1.7 mmol/L.
Fasting blood glucose level | 20 weeks
  Fasting blood glucose level will be measured in mmol/L. The healthy cut-off point of fasting blood glucose level is less than 6.1 mmol/L.
Body weight | 20 weeks
  Body weight will be assessed in kilograms.
Body height | Baseline
  Body height will be assessed in meters.
Body mass index | 20 weeks
  Body mass index (BMI) is derived from body weight in kilograms (kg) and body height in meters (m). BMI is expressed as kg/m^2.
Waist circumference | 20 weeks
  Waist circumference will be assessed in centimeters (cm). The healthy cut-off point of waist circumference for male is less than or equal to 90cm and for female less than or equal to 80cm.
Attitude and Beliefs about Cardiovascular Risk | 20 weeks
  Attitude and Beliefs about Cardiovascular Risk will be assessed using the Attitude and Beliefs about Cardiovascular Risk - Malay questionnaire. The overall score was calculated from all item scores by the domains. The higher the score, the higher the awareness and the readiness to change the behavior.
Physical activity level | 20 weeks
  The physical activity level will be assessed using the International Physical Activity Questionnaire. The intensity of self-reported physical activity lasting at least 10 minutes per bout was measured in metabolic equivalent (MET). The accumulated MET-minutes per week will be calculated to categorize into low, moderate (at least 600 MET-minutes per week) or high physical activity level (at least 3000 MET-minutes per week).
Medication Understanding and Taking Self-Efficacy | 20 weeks
  The Medication Understanding and Taking Self-Efficacy will be assessed using the Medication Understanding and Taking Self-Efficacy scale. The scores ranged from 8 to 32, with higher scores indicating greater levels of medication understanding.
Dietary intakes | 20 weeks
  The usual dietary intakes will be assessed using the short food frequency questionnaire. It provides details on daily intake of food groups.
Nutrient intakes | 20 weeks
  Nutrient intakes will be assessed using the 2-day 24-hour diet recalls. The participants will be asked about all details of the foods and beverages consumed in the past 24 hours, including the types of food, cooking methods, estimated portion size and brands. Nutrient intakes from 24-hour dietary recalls will be analyzed with Nutritionist Pro software (Axxya Systems, USA) to yield total energy, macronutrient and micronutrient intakes.
Stress level | 20 weeks
  The stress level will be assessed using the Perceived Stress Scale (PSS). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * 0-13 = low stress
  * 14-26 = moderate stress
  * 27-40 = high perceived stress
Smoking habit | 20 weeks
  Participants will be asked if they are non-smoker, past smoker or current smoker; how long have you been smoking; and how many cigarettes did/do you smoke per day?
Alcohol consumption | 20 weeks
  Participants will be asked if they are non-drinker, past drinker or current drinker; how long (years) have you been consuming alcohol?

CONTACTS AND LOCATIONS:
Overall Officials: Amutha Ramadas, PhD, Principal Investigator — Monash University Malaysia
Locations (1):
- Monash University, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim GP, Appalasamy JR, Ahmad B, Quek KF, Ramadas A. Peer-Led Digital Health Lifestyle Intervention in a Low-Income Community at Risk for Cardiovascular Disease (MYCardio-PEER): Mixed Methods Development and Process Evaluation Study. J Med Internet Res. 2025 Nov 12;27:e77063. doi: 10.2196/77063. PMID 41222971
- [Derived] Lim GP, Appalasamy JR, Ahmad B, Quek KF, Shaharuddin S, Ramadas A. Peer-led digital health lifestyle intervention for a low-income community at risk for cardiovascular diseases (MYCardio-PEER): a quasi-experimental study protocol. Prim Health Care Res Dev. 2025 Mar 3;26:e20. doi: 10.1017/S1463423625000192. PMID 40025749